CLINICAL TRIAL: NCT05108805
Title: Safety and Feasibility Study of Chimeric Antigen Receptor (CAR) T Cell Therapy With YESCARTA in the Outpatient Setting
Brief Title: Chimeric Antigen Receptor (CAR) T Cell Therapy With YESCARTA in the Outpatient Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Principal Investigator, Olalekan Oluwole, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC CTT 2109
Record Dates: First submitted 2021-10-29; First posted 2021-11-05 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Large B-cell Lymphoma; Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Blood Pressure; axicabtagene ciloleucel; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting (Experimental): Patients receive cyclophosphamide IV and fludarabine IV on days -5 to -3. Patients then receive YESCARTA IV for over 30 minutes on day 0 in the absence of disease progression of unacceptable toxicity.
  Interventions: Procedure: Telemedicine Visit; Procedure: Vital sign measurements; Procedure: Out-Patient Clinic Visit; Procedure: Blood pressure and pulse oximeter; Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Procedure: Telemedicine Visit — A remote telemedicine visit with audio and video, using the internet with a nurse practitioner (NP) located elsewhere. The participant and NP will activate the telemedicine App in their electronic device. Family will obtain vital signs (BP, heart rate (HR), respiration rate (RR), SPO2) and provide NP with the information. NP will also review the previous vital signs. Review of system questions are asked, and the answers given by subject recorded. Neurological assessment done, and ICE score calculated.
Procedure: Vital sign measurements — Participant and their family will record and measure vital signs using a wearable device and will place a call to the covering nurse practitioner to report the vital signs prior to reporting to the out patient visit.
Procedure: Out-Patient Clinic Visit — Physical exam and review of all available data
Procedure: Blood pressure and pulse oximeter — Participant and their family take their blood pressure and pulse oximeter
Biological: Axicabtagene Ciloleucel — Axicabtagene Ciloleuce given by IV
Drug: Cyclophosphamide — Given IV
  Other Names: Cyclophosphamide 500 mg/m^2/day; Cytoxan®
Drug: Fludarabine — Given IV
  Other Names: Fludarabine 30 mg/m^2/day; Fludara®

SUMMARY:
We hope to demonstrate that YESCARTA can be safely administered in the outpatient setting if we closely monitor subjects with physical exams, wearable devices, and telemedicine visits and only admit those who meet specified criteria

DETAILED DESCRIPTION:
Primary Objectives

* To explore the feasibility of treating subjects with YESCARTA in the outpatient setting and guide the development of a subsequent, larger study that will determine the tolerability and safety profile of YESCARTA in the outpatient setting.
* To determine the time to specific interventions post infusion and the number of subjects who remain outpatient through 72 hours, 7, 14, and 30 days.

Secondary Objectives:

* Identify risk factors that preclude outpatient administration, and to obtain clinical data that will guide the development of guidelines by which YESCARTA treatment in the outpatient setting can be done safely.
* Assess the impact of close monitoring with telemedicine and twice-daily physical exam on specific outcomes including CRS and ICANS in subjects treated with YESCARTA in the outpatient setting.
* Cumulative steroid exposure within 28 days post YESCARTA infusion.
* To calculate the estimated cost of YESCARTA administered in the outpatient setting.

Exploratory Objectives:

* Time from YESCARTA infusion to the following: fever, fever with neutropenia, fever without neutropenia.
* Time from fever to Tocilizumab, fever to ICU admission, fever to low BP, fever to IV Fluid, fever to vasopressor, fever to onset to arrhythmias and fever to hospitalization.
* Calculate modified Neutropenic Fever Symptom Burden (NFSB) score for days 1-3 for each subject. Appendix D
* Obtain subject reported outcomes measured by Subject-Reported Outcomes Measurement Information System (PROMIS; Appendix F) [16, 17]
* Feasibility of using wearable devices to monitor vital signs in the outpatient setting. Data collected are for research only

ELIGIBILITY:
Inclusion Criteria (before leukapheresis)

Age 18 years and above

Histologically proven large B cell lymphoma or transformed follicular lymphoma to DLBCL in relapse/refractory after two lines of therapies which included an anthracycline and CD20-targeted therapy.

Or

Chemotherapy refractory disease evidenced by lack of adequate response to first line therapy. This consists of either progressive disease as best response to first line therapy or stable disease as best response after 4 cycles of appropriate chemotherapy

Or

Refractory after autologous stem cell transplant (ASCT) at any time point

And

Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Adequate hematologic, hepatic, renal and cardiac function evidenced by:

* absolute neutrophil count (ANC) ≥1000/µL
* Platelet ≥ 75,000/ µL
* T-bilirubin ≤ 1.5 mg/dL
* Normal serum creatinine or creatinine clearance ≥ 60 mL/min/1.73 m2
* Cardiac ejection fraction ≥ 50%
* Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 5 times upper limit of normal (ULN).
* At least 1 measurable lesion
* Baseline oxygen saturation ≥92% on room air.
* Ability to stay at a distance which allows for subjects to come in and for specific interventions like antibiotics and tocilizumab to be started in 1 hour or less. This is approximately 30 miles of Vanderbilt.
* A caregiver who can be educated to operate equipment for vital signs monitoring.

Caregiver Eligibility:

Willingness to serve as a caregiver Ability to read, write and operate a phone Willingness to be taught to operate electronic device Willingness and ability to assist subject to wear electronic device such including patch, blood pressure machine, thermometer Pass caregiver assessment test

Subject and caregiver willing to be taught to operate an iPad or other electronic media for telemedicine, use wearable devices, and pass the caregiver competence test.

Exclusion Criteria:

History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years.

Known CD19 negative tumor.

History of Richter's transformation of chronic lymphocytic leukemia (CLL).

Autologous stem cell transplant with therapeutic intent within 6 weeks of planned YESCARTA infusion.

History of allogeneic stem cell transplantation.

Prior CAR therapy or other genetically modified T-cell therapy.

History of severe, immediate hypersensitivity reaction attributed to aminoglycosides.

Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the sponsor's medical monitor.

History of human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or hepatitis C infection. Subjects with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines or applicable country guidelines.

Presence of any in-dwelling line or drain (e.g., percutaneous nephrostomy tube, in-dwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters, such as a Port-a-Cath or Hickman catheter, are permitted.

Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases. Patients with treated secondary CNS involvement of lymphoma are allowed.

History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, progressive multifocal leukoencephalopathy, or any autoimmune disease with CNS involvement if it impairs ability to complete an effective and reliable neurological assessment.

Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.

History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrolment.

Requirement for urgent therapy due to tumor mass effects (e.g., blood vessel compression, bowel obstruction, or transmural gastric involvement).

Primary immunodeficiency.

Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.

Live vaccine ≤ 6 weeks prior to planned start of conditioning regimen.

History of severe immediate hypersensitivity reaction to any of the agents used in this study.

Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.

Subjects of both genders who are not willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy.

In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Must not have received immunomodulating agents including checkpoint inhibitors, Bruton tyrosine kinase (BTK) inhibitors, and Revlimid within 2 months or 5 half-lives whichever is shorter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olalekan Oluwole, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting: Patients receive cyclophosphamide IV and fludarabine IV on days -5 to -3. Patients then receive YESCARTA IV for over 30 minutes on day 0 in the absence of disease progression of unacceptable toxicity.
  Telemedicine Visit: A remote telemedicine visit with audio and video, using the internet with a nurse practitioner located elsewhere. The participant and NP will activate the telemedicine App in their electronic device. Family will obtain vital signs (BP, HR, RR, SPO2) and provide NP with the information. NP will also review the previous vital signs. Review of system questions are asked, and the answers given by subject recorded. Neurological assessment done, and ICE score calculated.
  Vital sign measurements: Participant and their family will record and measure vital signs using a wearable device and will place a call to the covering nurse practitioner to report the vital signs prior to reporting to the out patient visit.
  Out-Patient Clinic Visit: Physical exam and review of all available data
  Blood pressure and pulse oximeter: Participant and their family take their blood pressure and pulse oximeter
  Axicabtagene Ciloleucel: Axicabtagene Ciloleuce given by IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
Period: Overall Study
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Started | 25 (Number of patients that joined the study and underwent collection of T-cells for expansion.)
Completed | 20 (Number of patients that had successful T-cell expansion and was treated on study.)
Not Completed | 5
Not completed — T-cell expansion was not successful. | 5

BASELINE CHARACTERISTICS:
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Received YESCARTA
Description: The number of participants that received YESCARTA as outpatient therapy
Time Frame: Approximately 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Participants That Required Hospitalization at 72 Hours Post Infusion
Description: Number of subjects that were admitted to hospital at 72 hours post infusion
Time Frame: at 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 2

3. Primary Outcome: Participants That Required Hospitalization at 7 Days Post Infusion
Description: Number of subjects that were admitted to the hospital at 7 days post infusion
Time Frame: at 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 19

4. Primary Outcome: Participants That Required Hospitalization at 14 Days Post Infusion
Description: Number of subjects that were admitted to the hospital at 14 days post infusion
Time Frame: at 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 19

5. Primary Outcome: Participants That Required Hospitalization at 30 Days Post Infusion
Description: Number of subjects that were admitted to hospital at 30 days post infusion
Time Frame: at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 19

6. Secondary Outcome: Count of Risk Factors That Preclude Out-patient Administration of YESCARTA
Description: Reasons as to why a participant did not receive YESCARTA in the out-patient setting
Time Frame: Approximately 30 days
Population: This analysis includes all participants who consented to the study but did not receive YESCARTA as planned. Reasons the participants did not receive YESCARTA are listed.
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 5
Participants
  Death from progressive disease | 3
  Severe infection | 1
  Performance status change | 1

7. Secondary Outcome: Participants That Experienced Cytokine Release Syndrome Events
Description: Count of participants that had cytokine release syndrome events
Time Frame: Approximately 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 19

8. Secondary Outcome: Participants That Experienced Immune Effector Cell-associated Neurotoxicity Syndrome Events
Description: Count of participants that had an immune effector cell-associated neurotoxicity syndrome event
Time Frame: Approximately 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 8

9. Secondary Outcome: Incidence of Steroid Administration During YESCARTA
Description: Count of participants that were administered steroids during treatment
Time Frame: Approximately 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
Participants | 20

10. Secondary Outcome: Cost Per Patient of Administering YESCARTA in the Out-patient Setting
Description: Cost includes hospital clinic charges and CAR-T acquisition. It was pre-specified to report a single dollar amount that every participant was changed. The amount entered was the amount that each patient was charged. It was not planned to assess this amount separately for each participant.
Time Frame: Approximately 30 days
Population: This was the total cost per patient for administering Yescarta on study.
Measure: Number; unit: dollars
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
Number analyzed (Participants) | 20
dollars | 392,237.75

ADVERSE EVENTS:
Time Frame: From initiation of protocol-indicated treatment up to approximately 12 months.
Groups:
- YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting: Patients receive cyclophosphamide IV and fludarabine IV on days -5 to -3. Patients then receive YESCARTA IV for over 30 minutes on day 0 in the absence of disease progression of unacceptable toxicity.
  Telemedicine Visit: A remote telemedicine visit with audio and video, using the internet with a nurse practitioner located elsewhere. The participant and NP will activate the telemedicine App in their electronic device. Family will obtain vital signs (BP, HR, RR, SPO2) and provide NP with the information. NP will also review the previous vital signs. Review of system questions are asked, and the answers given by subject recorded. Neurological assessment done, and ICE score calculated.
  Vital sign measurements: Participant and their family will record and measure vital signs using a wearable device and will place a call to the covering nurse practitioner to report the vital signs prior to reporting to the out patient visit.
Arm/Group | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting
All-Cause Mortality (participants affected / at risk) | 6/25
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting (N=25)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | YESCARTA (Axicabtagene Ciloleucel) in the Outpatient Setting (N=25)
Anemia (Blood and lymphatic system disorders) | 3 (8)
White Blood Cell Decrease (Blood and lymphatic system disorders) | 3 (6)
Neutrophil Count Decrease (Investigations) | 10 (23)
Fatique (General disorders) | 8 (9)
Fever (General disorders) | 16 (19)
Platelet Count Decreased (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Hypotension (Vascular disorders) | 6 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Cognitive Disturbance (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 4 (6)
Headache (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 15 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT05108805/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT05108805/ICF_000.pdf